CLINICAL TRIAL: NCT01757834
Title: Efficacy of Shear Wave Ultrasound Elastography in Noninvasive Diagnosis of Thyroid Nodules
Brief Title: Shear Wave Ultrasound Elastography in Noninvasive Diagnosis of Thyroid Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Manjiri Dighe, Associate Professor of Radiology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 41443-EA; 1R21CA164112-01 (NIH)
Record Dates: First submitted 2012-12-12; First posted 2012-12-31 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Thyroid Nodule
Keywords: Thyroid Nodule; Thyroid Neoplasm; Differential Diagnosis; Elastography; Elasticity Imaging Technique; Sonoelastography
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SWUS Elastography (Experimental): This is a noninvasive technique using focused ultrasonic beams (pushing beams.) Several pushing beams at increasing depths are transmitted to generate a quasi-plane shear wave frame that propagates throughout the imaging area. After generating the shear wave, an ultrafast imaging sequence is performed to acquire successive raw radiofrequency dots at a very high frame rate (up to 20,000 per second). A tissue elasticity assessment can be derived from shear wave propagation speed. A color-coded image is displayed; softer tissue in blue and stiffer tissue in red. Quantitative information is delivered by drawing regions of interest on the thyroid and surrounding tissues which is the Elasticity Index expressed in kilo-Pascal (kPa). Due to the lack of manual compression and known value of the strength of pushing beam, SWUS gives an objective number to stiffness within the nodule.
  Interventions: Device: SWUS Elastography

INTERVENTIONS:
Device: SWUS Elastography
  Other Names: Aixplorer Ultrasound System (SuperSonic Imagine, Inc)

SUMMARY:
Shear wave ultrasound elastography is a new technique of finding the softness or hardness in tissue by applying a "push" generated by the machine. This technique will help in diagnosing malignancy in the thyroid gland without biopsy and avoiding biopsy in noncancerous nodules.

DETAILED DESCRIPTION:
Thyroid nodules are a common medical problem. With the wide use of various imaging modalities, incidentally detected thyroid nodules are becoming more common. However most of these nodules are benign with only a small proportion of 5-10% being malignant. With the increasing number of nodules detected, evaluation of these thyroid nodules presents a diagnostic challenge since the imaging modality used for evaluation at present, i.e., ultrasound (US) alone, has a low specificity of approximately 50-70%. In order to improve specificity to confidently diagnose malignancy in the thyroid nodule, a fine needle aspiration (FNA) biopsy is performed.

In recent years, US elastography has been shown to have high specificity of 90- 98% in various studies in differentiating between benign and malignant nodules. US elastography works on the principle of detecting the stiffness within a tissue by applying compression which can be manual compression or by generation of a remote radiation force by focused ultrasonic beams called as shear waves. Shear Wave Ultrasound (SWUS) elastography is an objective method of US elastography that detects the stiffness within the nodule since the strength of the shear wave generated is known and can be controlled. SWUS elastography has shown promise in being able to noninvasively diagnose papillary carcinoma in previous studies involving preoperative patients.

The investigators propose to perform a study to investigate the efficacy of SWUS elastography in diagnosing malignant thyroid nodules and noninvasively decreasing the number of FNAs performed by avoiding FNA in benign nodules. The Investigators will enroll patients with thyroid nodules before they undergo FNA biopsy or surgery. We also propose to compare routine US and SWUS elastography and their combined use in differentiating malignant from benign nodules. The investigators hypothesize that SWUS elastography can be used as a noninvasive screening tool, prior to an FNA, to screen out benign and malignant nodules with high level of confidence and reduce the number of biopsies in the future.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of thyroid nodule
* Referred for thyroid FNA or surgery

Exclusion Criteria:

* Minors; age <18
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Correlating stiffness from the SWUS elastography with indentometer and pathology findings | Up to 2 months. A one-time SWUS elastography will be performed on Day 1 within 2 months prior to the patients scheduled clinical FNA or surgery.
  SWUS elastography can provide an objective score of stiffness, i.e., the Elasticity Index.
  Stiffness from the SWUS elastography will be correlated with the elasticity measured with an indentometer to validate the Elasticity Index. The Elasticity Index will also be correlated with the histopathologic diagnosis. The sensitivity and specificity of the method for the diagnosis of malignancy will be assessed.

SECONDARY OUTCOMES:
Correlating SWUS findings with routine US findings | Up to 2 months. A one-time SWUS elastography will be performed on Day 1 within 2 months prior to the patients scheduled clinical FNA or surgery.
  The investigators will compare the SWUS findings to the routine US findings. This will help us develop criteria based on combined findings to decide if a thyroid nodule is suspicious enough to warrant a FNA biopsy. These criteria can then be used for future prospective studies.

CONTACTS AND LOCATIONS:
Overall Officials: Manjiri K. Dighe, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Frates MC, Benson CB, Charboneau JW, Cibas ES, Clark OH, Coleman BG, Cronan JJ, Doubilet PM, Evans DB, Goellner JR, Hay ID, Hertzberg BS, Intenzo CM, Jeffrey RB, Langer JE, Larsen PR, Mandel SJ, Middleton WD, Reading CC, Sherman SI, Tessler FN. Management of thyroid nodules detected at US: Society of Radiologists in Ultrasound consensus conference statement. Ultrasound Q. 2006 Dec;22(4):231-8; discussion 239-40. doi: 10.1097/01.ruq.0000226877.19937.a1. PMID 17146329
- [Background] Rago T, Santini F, Scutari M, Pinchera A, Vitti P. Elastography: new developments in ultrasound for predicting malignancy in thyroid nodules. J Clin Endocrinol Metab. 2007 Aug;92(8):2917-22. doi: 10.1210/jc.2007-0641. Epub 2007 May 29. PMID 17535993
- [Background] Gharib H, Goellner JR. Fine-needle aspiration biopsy of the thyroid: an appraisal. Ann Intern Med. 1993 Feb 15;118(4):282-9. doi: 10.7326/0003-4819-118-4-199302150-00007. PMID 8420446
- [Background] Lyshchik A, Higashi T, Asato R, Tanaka S, Ito J, Mai JJ, Pellot-Barakat C, Insana MF, Brill AB, Saga T, Hiraoka M, Togashi K. Thyroid gland tumor diagnosis at US elastography. Radiology. 2005 Oct;237(1):202-11. doi: 10.1148/radiol.2363041248. Epub 2005 Aug 18. PMID 16118150
- [Background] Dighe M, Bae U, Richardson ML, Dubinsky TJ, Minoshima S, Kim Y. Differential diagnosis of thyroid nodules with US elastography using carotid artery pulsation. Radiology. 2008 Aug;248(2):662-9. doi: 10.1148/radiol.2482071758. Epub 2008 Jun 6. PMID 18539888
- [Background] Bae U, Dighe M, Dubinsky T, Minoshima S, Shamdasani V, Kim Y. Ultrasound thyroid elastography using carotid artery pulsation: preliminary study. J Ultrasound Med. 2007 Jun;26(6):797-805. doi: 10.7863/jum.2007.26.6.797. PMID 17526611
- [Background] Utiger RD. The multiplicity of thyroid nodules and carcinomas. N Engl J Med. 2005 Jun 9;352(23):2376-8. doi: 10.1056/NEJMp058061. No abstract available. PMID 15944422
- [Background] Hegedus L. Clinical practice. The thyroid nodule. N Engl J Med. 2004 Oct 21;351(17):1764-71. doi: 10.1056/NEJMcp031436. No abstract available. PMID 15496625
- [Background] Papini E, Guglielmi R, Bianchini A, Crescenzi A, Taccogna S, Nardi F, Panunzi C, Rinaldi R, Toscano V, Pacella CM. Risk of malignancy in nonpalpable thyroid nodules: predictive value of ultrasound and color-Doppler features. J Clin Endocrinol Metab. 2002 May;87(5):1941-6. doi: 10.1210/jcem.87.5.8504. PMID 11994321
- [Background] American Thyroid Association (ATA) Guidelines Taskforce on Thyroid Nodules and Differentiated Thyroid Cancer; Cooper DS, Doherty GM, Haugen BR, Kloos RT, Lee SL, Mandel SJ, Mazzaferri EL, McIver B, Pacini F, Schlumberger M, Sherman SI, Steward DL, Tuttle RM. Revised American Thyroid Association management guidelines for patients with thyroid nodules and differentiated thyroid cancer. Thyroid. 2009 Nov;19(11):1167-214. doi: 10.1089/thy.2009.0110. PMID 19860577
- [Background] Gharib H, Papini E, Paschke R, Duick DS, Valcavi R, Hegedus L, Vitti P; AACE/AME/ETA Task Force on Thyroid Nodules. American Association of Clinical Endocrinologists, Associazione Medici Endocrinologi, and European Thyroid Association medical guidelines for clinical practice for the diagnosis and management of thyroid nodules. J Endocrinol Invest. 2010;33(5 Suppl):1-50. PMID 20543550
- [Background] Lyshchik A, Higashi T, Asato R, Tanaka S, Ito J, Hiraoka M, Brill AB, Saga T, Togashi K. Elastic moduli of thyroid tissues under compression. Ultrason Imaging. 2005 Apr;27(2):101-10. doi: 10.1177/016173460502700204. PMID 16231839
- [Background] Sebag F, Vaillant-Lombard J, Berbis J, Griset V, Henry JF, Petit P, Oliver C. Shear wave elastography: a new ultrasound imaging mode for the differential diagnosis of benign and malignant thyroid nodules. J Clin Endocrinol Metab. 2010 Dec;95(12):5281-8. doi: 10.1210/jc.2010-0766. Epub 2010 Sep 29. PMID 20881263
- [Background] Dighe M, Kim J, Luo S, Kim Y. Utility of the ultrasound elastographic systolic thyroid stiffness index in reducing fine-needle aspirations. J Ultrasound Med. 2010 Apr;29(4):565-74. doi: 10.7863/jum.2010.29.4.565. PMID 20375375
- [Background] Hong Y, Liu X, Li Z, Zhang X, Chen M, Luo Z. Real-time ultrasound elastography in the differential diagnosis of benign and malignant thyroid nodules. J Ultrasound Med. 2009 Jul;28(7):861-7. doi: 10.7863/jum.2009.28.7.861. PMID 19546328
- [Background] Tranquart F, Bleuzen A, Pierre-Renoult P, Chabrolle C, Sam Giao M, Lecomte P. [Elastosonography of thyroid lesions]. J Radiol. 2008 Jan;89(1 Pt 1):35-9. doi: 10.1016/s0221-0363(08)70367-6. French. PMID 18288024
- [Background] Luo S, Kim EH, Dighe M, Kim Y. Screening of thyroid nodules by ultrasound elastography using diastolic strain variation. Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:4420-3. doi: 10.1109/IEMBS.2009.5332744. PMID 19963828
- [Background] Itoh A, Ueno E, Tohno E, Kamma H, Takahashi H, Shiina T, Yamakawa M, Matsumura T. Breast disease: clinical application of US elastography for diagnosis. Radiology. 2006 May;239(2):341-50. doi: 10.1148/radiol.2391041676. Epub 2006 Feb 16. PMID 16484352
- [Background] Luo S, Kim EH, Dighe M, Kim Y. Thyroid nodule classification using ultrasound elastography via linear discriminant analysis. Ultrasonics. 2011 May;51(4):425-31. doi: 10.1016/j.ultras.2010.11.008. Epub 2010 Nov 27. PMID 21163507
- [Background] Erkamp RQ, Wiggins P, Skovoroda AR, Emelianov SY, O'Donnell M. Measuring the elastic modulus of small tissue samples. Ultrason Imaging. 1998 Jan;20(1):17-28. doi: 10.1177/016173469802000102. PMID 9664648
- [Background] Parker KJ, Huang SR, Musulin RA, Lerner RM. Tissue response to mechanical vibrations for "sonoelasticity imaging". Ultrasound Med Biol. 1990;16(3):241-6. doi: 10.1016/0301-5629(90)90003-u. PMID 2194336
- [Background] Iannuccilli JD, Cronan JJ, Monchik JM. Risk for malignancy of thyroid nodules as assessed by sonographic criteria: the need for biopsy. J Ultrasound Med. 2004 Nov;23(11):1455-64. doi: 10.7863/jum.2004.23.11.1455. PMID 15498910